CLINICAL TRIAL: NCT01403870
Title: Post Market Study of the Electrophysiological Course of Low Back Pain Using CERSR Technology
Status: Terminated | Type: Observational
Why Stopped: Company no longer has funding for the study.
Sponsor: Verium Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011-001
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Low Back Pain
Keywords: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Low Back Pain Subjects: Subjects who have low back pain at the time of the study, and wish to receive physical therapy to reduce their low back pain.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — The physician will complete a physical exam as well as analyze a completed CERSR scan study to determine the root cause of the low back pain. The physician will then prescribe a targeted physical therapy regime to address the cause of the low back pain.

SUMMARY:
The purpose of this research study is:

1. to measure with CERSR® (Computerized Electrophysiological Reconstruction of the Spinal Regions) the electrical signals made by the muscles in the lower back during the treatment of the low back pain, and
2. to study the changes which take place in these muscles with treatment. The device is non-invasive which means nothing is put into your body. The CERSR® pad is an adhesive (sticky) array (ordered rows) of electrodes.

The investigators hope to find information about the quality of the muscles' electrical signals in reaction to injury causing back pain, which will improve understanding of the nature of back pain and back injury. The investigators also hope to improve treatment by creating a simple test, which will tell us objectively (through computerized measurement) whether the treatment is helping.

DETAILED DESCRIPTION:
Verium Diagnostics, Inc., has developed a non-invasive device to aid the Physician in the diagnosis of muscle disease and muscle dysfunction. CERSR® (Computerized Electrophysiological Reconstruction of the Spinal Regions), is a non-invasive diagnostic procedure to "Monitor and display the bioelectric signals produced by muscles to aid in the diagnosis and prognosis of muscular disease and dysfunction." The technology captures electrophysiological data and introduces it into reconstructive algorithms similar to those used in Magnetic Resonance Imaging (MRI) and Positron Emission Tomography (PET). The technology has been developed to overcome the problems associated with surface EMG technology. SEMG is limited by a resolution problem related to distance separating the electrodes from the muscle (subcutaneous thickness), number and location of electrodes applied, as well as limits on the minimum distance separating the electrodes, and on cross interference between electrode pairs.

The CERSR® scan is a procedure which monitors and displays the bioelectric signals produced by the paraspinal neuromuscular system. A disposable large surface array of 63 sensors (7 across x 9 down) is placed on the back, using T7 & L4 as landmarks. The array is connected to a computer that is calibrated to read the neuromuscular activity covered by the electrode grid. Three scans are captured by the software in each of three different positions: A) Standing relaxed with arms at sides; B) Body flexed at the hips to a 20° angle and C) Standing with the arms outstretched in front holding a 3 lb. weight in each hand. The electrophysiological information is processed with a highly proprietary imaging software program. The scans collect 1,953 bioelectric signals generated by the 96 muscles and 60 nerves that make up the paraspinal neuromuscular system, and within two seconds results in an image that reflects the muscle recruitment pattern of the paraspinal region.

The reconstructed physiological data are presented to the physician in a multitude of readily interpreted images of the lower back with data-inclusive reports. The software translates the registered activity into a color grid, with slight activity represented by blue and red signifying intense contractility. Normal back musculature activity is characterized by a centralized, symmetrical image pattern. Abnormal low back musculature activity is characterized by non-symmetric and/or multi-focal images signifying abnormal muscular activity. In addition to the images, which reflect the recruitment of muscle associated with the bioelectric signals, the software has been developed to calculate a Root Mean Square voltage (RMS) between each electrode as well as a mean for the entire electrode array. This Power Value increases as the bioelectric signals increase, and decreases as the bioelectric signals decrease. The images and associated Power Values can aid the Physician in the diagnosis and prognosis of muscle disease and dysfunction.

A previous clinical pilot study of the CERSR® technology using 201 subjects with and without low back pain1 and an analysis of data gather by CERSR® methodology in a trial of 161 healthy volunteers and 44 acute low back pain patients2, have demonstrated that:

1. Persons with acute onset of low back pain have abnormal EMG signals, which can be reliably mapped using CERSR® technology 1.
2. The scan results generated by CERSR for a normal subject (no low back pain), differs from the scan results for a not normal subject (low back pain present) 1,2,
3. The abnormal EMG signals will return to normal as medical treatment results in resolution of pain and dysfunction 1.
4. Root Mean Square (RMS) values from subjects with low back pain are different than RMS values from normal pain-free subjects 1,2.

The purpose of the proposed study is to assess the efficacy of using the CERSR® imagining technology to 1) identify individuals with low back pain, 2) to investigate whether the use of the CERSR® technology can successfully aid the physician to direct a therapeutic regimen that can provide relief to treated subjects, and 3) to demonstrate that the CERSR® technology can be used to track and document progress and success of the directed therapy regime. It is believed that the use of the CERSR® methodology, and the resulting physician directed therapy being investigated in this study, will result in significant cost savings through reduced diagnostic procedure and medical treatment related costs, and shorter treatment lengths. CERSR® data from serial scanning may also be able to be compared to baseline CERSR® results to assist the Physician in determining Maximum Medical Improvements.

The purpose of this research study is

1. to measure with CERSR® (Computerized Electrophysiological Reconstruction of the Spinal Regions) the electrical signals made by the muscles in the lower back during the treatment of the low back pain, and
2. to study the changes which take place in these muscles with treatment. The device is non-invasive which means nothing is put into your body. The CERSR® pad is an adhesive (sticky) array (ordered rows) of electrodes.

The investigators hope to find information about the quality of the muscles' electrical signals in reaction to injury causing back pain, which will improve understanding of the nature of back pain and back injury. The investigators also hope to improve treatment by creating a simple test, which will tell us objectively (through computerized measurement) whether the treatment is helping.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female who have VHN medical coverage.
2. Between the ages of 18 and 70

Exclusion Criteria:

1. Low back pain due to fracture, tumor, infection, cauda equina, severe neurological deficit
2. Pregnant
3. Sensitivity to isopropyl alcohol used to prepare the low back surface
4. Inability to complete the required collection positions for the CERSR® scan
5. Inability or unwillingness to adhere to the protocol and follow-up schedule
6. Anyone under care of a physician for active liability or workman compensation cases.
7. Anyone who has had an open spinal procedure in the last three months.
8. Anyone who has undergone spine injections within the last two months.
9. Anyone who is currently undergoing physical therapy or chiropractic treatments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Test subjects will be recruited from individuals who are currently have Volusia Health Network (VHN) medical coverage.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-04

PRIMARY OUTCOMES:
Change from Baseline in Pain Visual Analog Scale | Upon enrollment (day 1 - baseline) and four weeks and eight weeks
  The subjects will complete a form indicating their pain level upon enrollment. Subjects will then be scanned again at four weeks and at eight weeks. At the time of the scan subjects will also be asked to complete a follow up VAS. Upon completion of the study the change in the VAS scores will be analyzed.

SECONDARY OUTCOMES:
Change from Baseline Oswestry Disability Index (ODI) | Upon enrollment (day 1 - baseline) and at four weeks and at eight weeks
  The subjects will complete the Oswestry Disability Index (ODI) upon enrollment. Subjects will then be scanned again at four weeks and at eight weeks. At the time of the scan subjects will also be asked to complete a follow up ODI. Upon completion of the study the change in the ODI scores will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gillespy, M.D., Principal Investigator — Orthopaedic Clinic of Daytona Beach
Locations (1):
- Orthopaedic Clinic of Daytona Beach, Daytona Beach, Florida, United States

REFERENCES:
- [Result] Finneran MT, Mazanec D, Marsolais ME, Marsolais EB, Pease WS. Large-array surface electromyography in low back pain: a pilot study. Spine (Phila Pa 1976). 2003 Jul 1;28(13):1447-54. doi: 10.1097/01.BRS.0000067565.16832.B9. PMID 12838104